CLINICAL TRIAL: NCT05543902
Title: The Effects of the Breastfeeding Problems Management Model (BPMM) on Breastfeeding Problems, Breastfeeding Motivation and Breastfeeding Success: A Randomized Clinical Trial
Brief Title: The Effects of the Breastfeeding Problems Management Model on Breastfeeding Problems, Motivation and Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra ÇERÇER, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-25
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Counselling
Keywords: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Breastfeeding Problems Management Model (BPMM) (Experimental): The women in the intervention group were provided with nursing interventions according to the BPMM by the researcher. LATCH (pre-test) was administered before discharge from the hospital; women were given the education booklet; and their contact information was recorded. After discharge from the hospital, the women were called by phone in the 1st, 2nd, and 6th weeks, BES was read, and the scale was filled in by the researcher based on the women's responses. Women who were found to experience breastfeeding problems in these phone calls were provided with consultancy and home visits. In the 8th week, home visits were done and the education was repeated. The women were administered the BES, LATCH (post-test), and BMS.
  Interventions: Behavioral: Breastfeeding Problems Management Model (BPMM)
- No Intervention: Standard care group (No Intervention): The women in standard care group were not provided with any interventions by the researcher. They were provided with standard care at the hospital. Before discharge from the hospital, the LATCH (pre-test) was administered and women's contact information was recorded. After discharge from the hospital, the women were called by phone in the 1st, 2nd, and 6th weeks. BES were read on the phone, and the scale was filled in by the researcher based on the women's responses. Home visits were performed in the 8th week, and the women were administered the BES, LATCH (post-test), and BMS

INTERVENTIONS:
Behavioral: Breastfeeding Problems Management Model (BPMM) — The BPMM was composed of interventions with the leadership of a nurse and included topics of the early postpartum period; postpartum 1st, 2nd, 6th, and 8th weeks; increasing breastfeeding motivation and breastfeeding success; and preventing and eliminating breastfeeding problems. The components of the model included meeting women face-to-face, giving education using a booklet, providing breastfeeding consultancy on the phone, and home visits.
  Arms: Intervention group: Breastfeeding Problems Management Model (BPMM)

SUMMARY:
This randomized controlled interventional study was conducted with 50 women (25 intervention and 25 control). While the intervention group received an eight-week postpartum education and care according to the Breastfeeding Problems Management Model (BPMM) under the leadership of a nurse, the control group received routine care. CONSORT checklist was used to report the study.The women in the intervention group were provided with nursing interventions according to the BPMM by the researcher. The women in standard care group were not provided with any interventions by the researcher.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled trial to determine the effects of the Breastfeeding Problems Management Model (BPMM) on breastfeeding problems, breastfeeding motivation and breastfeeding success.

Research hypotheses H0: Mothers in the intervention and control group H01: Demonstrate no differences in terms of their "LATCH Assessment Tool" total mean scores.

H02: Demonstrate no differences in terms of their "Breastfeeding Motivation Scale" total mean scores.

H03: Demonstrate no differences in terms of their "Breastfeeding Experience Scale" total mean scores.

H1: Mothers in the intervention and control group H11: Demonstrate differences in terms of their "LATCH Assessment Tool" total mean scores.

H12: Demonstrate differences in terms of their "Breastfeeding Motivation Scale" total mean scores.

H13: Demonstrate differences in terms of their "Breastfeeding Experience Scale" total mean scores.

This study was conducted in the Obstetrics and Gynecology Clinic at Adana City Training and Research Hospital affiliated with the T.R. Ministry of Health between 01/06/2020 and 01/04/2022. The target population of the study included women who had a vaginal delivery at Adana City Training and Research Hospital affiliated with the T.R. Ministry of Health. The sample of the study was women who had vaginal delivery in the related hospital between 01/06/2020 and 01/04/2022, who met the research criteria, and who agreed to participate in the study.

Power analysis was performed after data were collected from 20 women who had a vaginal delivery (10 intervention, 10 control) for the calculation of the sample size. Power analysis conducted using values obtained from the pilot implementation via the G*Power 3.0.10, for 4 repeat models with 80% Power and 5% margin of error, indicated that at least 40 samples were adequate for 2 groups (n1:20; n2:20). Due to the probability of women's leaving the study during their follow-ups, the study included 50 women: 25 intervention and 25 control group participants.

Data were collected through the "Personal Information Form", the "Breastfeeding Experience Scale", the "LATCH Assessment Tool", and the "Breastfeeding Motivation Scale (for Primiparous Mothers)".

The study formed the "Breastfeeding Problems Management Model (BPMM)", and the nursing interventions in the intervention group were done based on this model.The BPMM was composed of interventions with the leadership of a nurse and included topics of the early postpartum period; postpartum 1st, 2nd, 6th, and 8th weeks; increasing breastfeeding motivation and breastfeeding success; and preventing and eliminating breastfeeding problems. The components of the model included meeting women face-to-face, giving education using a booklet, providing breastfeeding consultancy on the phone, and home visits.

The women in the intervention group were provided with nursing interventions according to the BPMM by the researcher. LATCH (pre-test) was administered before discharge from the hospital; women were given the education booklet; and their contact information was recorded. After discharge from the hospital, the women were called by phone in the 1st, 2nd, and 6th weeks, BES was read, and the scale was filled in by the researcher based on the women's responses. Women who were found to experience breastfeeding problems in these phone calls were provided with consultancy and home visits. In the 8th week, home visits were done and the education was repeated. The women were administered the BES, LATCH (post-test), and BMS.

The women in control group were not provided with any interventions by the researcher. They were provided with standard care at the hospital. Before discharge from the hospital, the LATCH (pre-test) was administered and women's contact information was recorded. After discharge from the hospital, the women were called by phone in the 1st, 2nd, and 6th weeks. BES were read on the phone, and the scale was filled in by the researcher based on the women's responses. Home visits were performed in the 8th week, and the women were administered the BES, LATCH (post-test), and BMS.

ELIGIBILITY:
Inclusion Criteria:

1. being aged between 18 and 35
2. having vaginal delivery in the 37th gestational week or later
3. being primiparous
4. having a single and healthy fetus
5. having graduated at least from a primary school
6. living in Adana city center
7. being able to communicate on the phone.

Exclusion Criteria:

1. having no high-risk pregnancy
2. having no medical diseases preventing breastfeeding
3. having no communication problems
4. having no psychiatric diseases
5. not being a health professional
6. having no health professional relatives to provide support in the postpartum care.

Criteria for being excluded from the study:

1. admission of the newborn to the intensive care
2. development of postpartum psychological problems in the mother (maternity blues, depression)
3. mother's changing city during postpartum follow-ups.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Experience Scale (BES) | Change in breastfeeding problems by 1st, 2nd, 6th and 8th weeks
  The original scale is responded on a 5-point scale and is composed of 2 parts, 5 sub-scales, and 30 items. Turkish reliability and validity of the scale were performed by Uyanık and Çeber Turfan in 2019, and Cronbach's alpha coefficient was found 0.776. Scores to be obtained from the scale range between 18 and 90, with higher scores indicating higher severity of breastfeeding problems. BES was reported to be a valid tool for the Turkish Society.

SECONDARY OUTCOMES:
The LATCH Assessment Tool | Change in 1th and 8th weeks breastfeeding succes level.
  The LATCH Assessment Tool was developed by Jensen et al. in 1994. Reliability analysis of the tool was performed by Adams and Hewel in 1997. Turkish reliability and validity were performed by Yenal and Okumuş in 2001 and Cronbach's alpha coefficient was reported 0.95, indicating the reliability of the scale. The LATCH is composed of 5 criteria that enable a rapid and easy assessment: L: Latch on breast, A: Audible swallowing, T: Type of nipple, C: Comfortbreast/nipple, H: Hold. Each item is scored between 0 and 2, and the scores to be obtained from the scale range between 0 and 10. Higher scores indicate successful breastfeeding.

OTHER OUTCOMES:
The Breastfeeding Motivation Scale (BMS) | change in breastfeeding motivation level at eight weeks
  Turkish reliability and validity of the scale were performed by Mızrak. BMS for primiparous women is composed of 23 items and 5 sub-scales. The scale is rated on a 4-point Likert scale (1: I strongly disagree, 4: I strongly agree). The scale has no total score; the average of the sub-scale scores is calculated. Higher scores indicate increased motivation representing that sub-scale. Mızrak administered the scale to mothers in the 8th week. Cronbach's alpha value was found 0.887 in the scale for primiparous mothers, and Cronbach's alpha values were found between 0.658 and 0.879 for the sub-scales. Turkish version of the BMS was found to be a valid and reliable tool for determining mothers' breastfeeding motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra ÇERÇER, PhD, Principal Investigator — Cukurova University; Evşen NAZİK, Prof. Dr., Study Director — Cukurova University
Locations (1):
- Cukurova Unıversity, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucas R, Zhang Y, Walsh SJ, Evans H, Young E, Starkweather A. Efficacy of a Breastfeeding Pain Self-Management Intervention: A Pilot Randomized Controlled Trial. Nurs Res. 2019 Mar/Apr;68(2):E1-E10. doi: 10.1097/NNR.0000000000000336. PMID 30829925
- [Background] Lucas R, Bernier K, Perry M, Evans H, Ramesh D, Young E, Walsh S, Starkweather A. Promoting self-management of breast and nipple pain in breastfeeding women: Protocol of a pilot randomized controlled trial. Res Nurs Health. 2019 Jun;42(3):176-188. doi: 10.1002/nur.21938. Epub 2019 Mar 5. PMID 30835887
- [Background] Mizrak Sahin B, Ozerdogan N, Ozdamar K, Gursoy E. Factors affecting breastfeeding motivation in primiparious mothers: An application of breastfeeding motivation scale based on self-determination theory. Health Care Women Int. 2019 Jun;40(6):637-652. doi: 10.1080/07399332.2018.1526289. Epub 2019 May 29. PMID 31140955
- [Derived] Cercer Z, Nazik E Dr. The effects of the breastfeeding problems management model on breastfeeding problems, breastfeeding motivation and breastfeeding success: A randomized controlled trial. J Pediatr Nurs. 2023 Nov-Dec;73:e116-e124. doi: 10.1016/j.pedn.2023.07.021. Epub 2023 Aug 6. PMID 37550129